CLINICAL TRIAL: NCT03617419
Title: Evaluation of Feasibility and Accuracy of Assisted Fetal Heart Rate (FHR) Feature of the GE Vscan Access R2 Ultrasound System
Brief Title: Vscan Access R2 Feasibility Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 110.05-2017-GES-0001
Record Dates: First submitted 2018-03-01; First posted 2018-08-06 (Actual); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Gather Feasibility Data and User Feedback on Use of a Device in Vivo on Pregnant Volunteers in Their 2nd and 3rd Trimester

STUDY DESIGN:
Intervention Model Description: This study is being done to evaluate and gather feasibility data and user feedback on the use of the Vscan Access R2 device in vivo on pregnant volunteers in their 2nd and 3rd Trimester. The study will be conducted in two parts, including an initial pilot for determination of parameters (Part 1) and continued testing (Part 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- VScan Access R2 Ultrasound System (Other): Pre-market: Vscan Access R2 Ultrasound System
  The following post-market products will be used on label:
  GE Corometrics 170 Series Fetal Monitor - as a reference for value of fetal heart rate GE Voluson P8 Ultrasound System - for verification of fetal location during measurement
  Interventions: Device: GE VScan Access R2 Ultrasound System; Device: GE Corometrics 170 Series Fetal Monitor

INTERVENTIONS:
Device: GE VScan Access R2 Ultrasound System — A diagnostic ultrasound imaging system manufactured by the study Sponsor.
Device: GE Corometrics 170 Series Fetal Monitor — A reference device to record a continuous fetal heart rate.
Device: GE Corometrics 170 Series Fetal Monitor — A reference device for verification of scanning the fetal heart.

SUMMARY:
This study is being done to evaluate if the Vscan Access R2 Ultrasound System can measure Fetal Heart Rate (FHR) in humans when compared against a reference device (GE Corometrics 170 Series Fetal Monitor), and to gather feedback from device operators on the usability of the device.

DETAILED DESCRIPTION:
This study is being done to evaluate whether the Vscan Access R2 Ultrasound System Assisted FHR phantom testing conclusions can be extrapolated onto human fetal heart rate measurements, where CTG (GE Corometrics 170 Series Fetal Monitor) is to provide a reference value. It should be noted that the Vscan Access R2 Ultrasound System with Assisted FHR has a different intended use than CTG (momentary FHR value versus continuous monitoring of FHR patterns and trends) and this aspect is out of scope of this research.

Usability data will be gathered for further user experience optimization.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or older at the time of consent;
2. By self-report, are in the 2nd or 3rd trimester of pregnancy;
3. Able and willing to provide written informed consent for participation;
4. Provide a completed Healthcare Verification Form which confirms the subject has received at least one diagnostic ultrasound during this pregnancy and has an uncomplicated pregnancy.

Exclusion Criteria:

1. Are direct employees/contractors of General Electric (GE);
2. Are potentially put at additional risk by participating, in the opinion of study staff;
3. Twin pregnancies identified in patient medical history.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study of pregnant volunteers
Enrollment: 16 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GE Healthcare - Milwaukee County Research Park, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VScan Access R2 Ultrasound System: Pre-market: Vscan Access R2 Ultrasound System
  The following post-market products will be used on label:
  GE Corometrics 170 Series Fetal Monitor - as a reference for value of fetal heart rate GE Voluson P8 Ultrasound System - for verification of fetal location during measurement
  GE VScan Access R2 Ultrasound System: A diagnostic ultrasound imaging system manufactured by the study Sponsor.
  GE Corometrics 170 Series Fetal Monitor: A reference device to record a continuous fetal heart rate.
  GE Corometrics 170 Series Fetal Monitor: A reference device for verification of scanning the fetal heart.
Period: Part 1
Arm/Group | VScan Access R2 Ultrasound System
Started | 2
Completed | 2
Not Completed | 0
Period: Part 2
Arm/Group | VScan Access R2 Ultrasound System
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data and results collected/analyzed for participants in active study phase (2). Pilot participant data not collected per study Protocol.
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Trimester (2nd or 3rd) [Count of Participants; unit: Participants]
  2nd Trimester of Pregnancy | 8
  3rd Trimester of Pregnancy | 6

OUTCOME MEASURES:

1. Primary Outcome: Difference in Fetal Heart Rate as Measured by VScan Access R2 and Corometrics
Description: Absolute difference and variance in fetal heart rate (in BPM) measured using VScan Access R2 and Corometrics
Time Frame: 1 day - Up to 45 minutes of total scan time
Measure: Mean (Standard Deviation); unit: Beats Per Minute (BPM)
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 14
Beats Per Minute (BPM) | 4.2 (4.13)

2. Secondary Outcome: GE Voluson P8 Confirmation of Visualization of Fetal Heart With Yes/No Answer Per Subject
Description: Visualization of fetal heart as acquired from the GE Voluson P8 to verify that the fetal heart was correctly identified during the image acquisition using Vscan Access R2. This is gathered through a Yes/No confirmation by device operator as to whether it was the fetal heart being scanned (once for each subject).
Time Frame: 1 day - Up to 45 minutes of total scan time (5 minutes for this specific measurement)
Population: Subjects in Part 1 (2) and Part 2 (14)
Measure: Number; unit: "Yes" responses
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 16
"Yes" responses | 16

3. Other Pre Specified Outcome: Number of Adverse Events (AE/SAE) Reported During Study
Description: Summary of type and number of AEs, SAEs reported/recorded during course
Time Frame: Collected from the time subject signs informed consent form to the time of completion of subject's scan session, estimated up to 4 hours
Measure: Number; unit: AEs / SAEs Reported
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 16
AEs / SAEs Reported | 0

4. Other Pre Specified Outcome: Number of Scan Operators Who Completed Surveys Regarding Usability of Vscan Access R2 Device
Description: Series of nine questions regarding usability, ease of use, and workflow
Time Frame: 10 minute survey completed by scan operators upon completion their participation (only one day per user)
Population: Device Operators
Measure: Number; unit: Completed Usability Surveys
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 9
Completed Usability Surveys | 9

5. Other Pre Specified Outcome: Number of Device Issues/Complaints Reported by Site
Description: Device Issues, Complaints, and Malfunctions will be reported in a table (type and number)
Time Frame: Three weeks (estimated study duration)
Measure: Number; unit: Device Malfunctions
Arm/Group | VScan Access R2 Ultrasound System
Number analyzed (Participants) | 16
Device Malfunctions | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection period for duration of study scanning (~ one week).
Description: Subject were monitored for AEs, SAEs, and UADEs during their study exams, until they exited the exam area. Procedures were conducted during a single visit (about one hour for each subject).
Arm/Group | VScan Access R2 Ultrasound System
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03617419/Prot_SAP_000.pdf